CLINICAL TRIAL: NCT02965521
Title: Survivor Choices for Eating and Drinking - Colorectal Cancer
Acronym: SUCCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 164511; NCI-2017-01381 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Rectal Cancer; ColoRectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Masking Description: Statistician who analyzes the data will be masked to intervention/control status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be given print material on diet for cancer survivors and access to a web-based dietary intervention with text messaging for 12 weeks.
  Interventions: Behavioral: Website and text messages
- Control (No Intervention): Participants randomized to the control arm will receive print materials on diet for cancer survivors. After completion of their 12-week follow-up assessments, control participants will be given access to the web-based dietary intervention with text messaging for 12 weeks.

INTERVENTIONS:
Behavioral: Website and text messages — Participants receive a personalized diet report, access to a digital health dietary intervention, and text messages for 12 weeks.
  Arms: Intervention

SUMMARY:
Epidemiologic data suggest that a Western dietary pattern after diagnosis of colorectal cancer increases risk of disease recurrence and death. High intake of red and processed meat, dairy, refined grains, and sweets/desserts characterize a 'Western dietary pattern'. This study aims to translate the epidemiologic findings into a patient-centered, web-based dietary intervention with text messaging to inform and modify users' dietary choices. The investigators' specific aims are to: 1) Develop a web-based dietary intervention with text messaging for colorectal cancer survivors; and 2) Conduct a 12-week pilot randomized controlled trial to determine the acceptability and feasibility of the dietary intervention among 50 colorectal cancer survivors. All participants will receive standard of care print materials regarding diet following a colorectal cancer diagnosis. Participants in the intervention group will also receive access to a web-based dietary intervention with text messaging for 12 weeks. This study will generate preliminary data on the effect of the intervention on dietary choices among colorectal cancer survivors for future studies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with colon or rectal adenocarcinoma
* completed standard cytotoxic chemotherapy prior to enrollment, if medically indicated
* considered disease-free or have stable disease at baseline
* able to speak and read English
* access to a mobile phone with Internet and text messaging capabilities
* able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the Internet

Exclusion Criteria:

Individuals who are already meeting four or more of the six target dietary behaviors will be excluded:

* ≥5 servings/day of fruits & vegetables
* ≥3 servings/day of whole grains
* ≥2 servings/week of fish
* no processed meat
* no sugar-sweetened beverages
* ≤1 alcoholic drink/d for women and ≤2 alcoholic drinks/d for men.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Adherence | 12-weeks
  Frequency of logging on to website and responding to text messages

SECONDARY OUTCOMES:
Dietary change assessed via diet records | 12-weeks
  Change in consuming vegetables, whole grains, fish, processed meat, sugar-sweetened beverages, and alcohol
Quality-of-life (EORTC C30) | 12-weeks
  Change in quality-of-life
Colorectal cancer-specific quality-of-life (EORTC C30 CR29) | 12-weeks
  Change in colorectal cancer-specific quality-of-life
Change in body mass index | 12-weeks
  Change in objectively measured BMI
Change in waist circumference | 12-weeks
  Change in objectively measured waist circumference
Change in fasting blood lipids | 12-weeks
  Change in fasting blood lipids
Change in fasting glucose | 12-weeks
  Change in fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Erin Van Blarigan, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Wang L, Langlais C, Kenfield SA, Van Loon K, Laffan A, Atreya CE, Chan JM, Zhang L, Allen IE, Miaskowski C, Fukuoka Y, Meyerhardt JA, Venook AP, Van Blarigan EL. Quality of life among colorectal cancer survivors participating in a pilot randomized controlled trial of a web-based dietary intervention with text messages. Support Care Cancer. 2023 Feb 10;31(3):155. doi: 10.1007/s00520-023-07620-x. PMID 36763183
- [Derived] Van Blarigan EL, Kenfield SA, Chan JM, Van Loon K, Paciorek A, Zhang L, Chan H, Savoie MB, Bocobo AG, Liu VN, Wong LX, Laffan A, Atreya CE, Miaskowski C, Fukuoka Y, Meyerhardt JA, Venook AP. Feasibility and Acceptability of a Web-Based Dietary Intervention with Text Messages for Colorectal Cancer: A Randomized Pilot Trial. Cancer Epidemiol Biomarkers Prev. 2020 Apr;29(4):752-760. doi: 10.1158/1055-9965.EPI-19-0840. Epub 2020 Jan 15. PMID 31941707